CLINICAL TRIAL: NCT04409756
Title: Validity and Reliability of the Turkish Version of the Shoulder Rating Questionnaire
Brief Title: Shoulder Rating Questionnaire in Turkish
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Betül Tepeli (Other)
Collaborators: Ufuk University (Other)
Responsible Party: Sponsor-Investigator, Betül Tepeli, Department of Physical Medicine And Rehabilitation, Private Balkan Hospital,Principal Investigator,, Namik Kemal University
Organization: Namik Kemal University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20181106/4
Record Dates: First submitted 2020-05-25; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Shoulder Pain
Keywords: Disability Evaluation; Shoulder Pain; Shoulder Validation Studies; Outcome measures
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- postassessment of the SRQ-T test (Other): the SRQ -T will be obtained to all patients three days after the first assessment
  Interventions: Other: shoulder rating questionnaire

INTERVENTIONS:
Other: shoulder rating questionnaire — to investigate reliability of turkish version of shoulder rating questionnaire

SUMMARY:
The purpose of this study is to determine the Turkish version of the Shoulder Rating Questionnaire (SRQ) and assign reliability and validity in Turkish patients.

DETAILED DESCRIPTION:
Shoulder pain is one of the common musculoskeletal disorders. A self- administered patient-based questionnaire has an important role for evaluate shoulder disabilities and also it is helpful for assess the treatment success.The purpose of this study is to determine the Turkish version of the Shoulder Rating Questionnaire (SRQ) and assign reliability and validity in Turkish patients.The Turkish version of the Shoulder Rating Questionnaire (SRQ-T) will be applied to patients after translation from English into Turkish. 122 patients will be participate to the study. Patients who were over 18 years with various shoulder pain complaints will be included into the study. The patients with mixed-type pain, cancer pain, headache, substance abuse, severe depression and fibromyalgia syndrome will be excluded. The musculoskeletal and neurological examinations of the patients will be performed. The Turkish version of the Shoulder Rating Questionnaire (SRQ-T) and Disabilities of arm, shoulder, hands-T (DASH-T) will be applied to all patients.

SRQ-T and DASH-T will be collected in two sessions with at last three days between the sessions for pre-assessment and post-assessment. Reliability of SRQ-T questionnaire will be tested by internal consistency and test-retest reliability. Internal consistency will be evaluated by determining intraclass correlation coefficient (ICC) with 95% confidence interval, ranged between 0 and 1.

To determine the internal consistency of the five domains of SRQ-T, Cronbach's alfa coefficient will be computed for both pre- and post-assessment of the questionnaire. The test-retest method with Wilcoxon Signed Rank Test will be used to determine reliability of SRQ-T and its domains. Then, Spearman correlation coefficients will be used to assess the discriminant validity of SRQ-T for evaluation of shoulder pain. The Spearman correlation coefficient score more than 0.70 will be accepted for reliability

ELIGIBILITY:
Inclusion Criteria:

* Patients who were over 18 years with various shoulder pain complaints

Exclusion Criteria:

* The patients with mixed-type pain, cancer pain, headache, substance abuse, severe depression and fibromyalgia syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
reliability of SRQ-T questionnaire | through study completion, an average of 1 month
  Reliability of SRQ-T questionnaire will be tested by internal consistency and test-retest reliability. Internal consistency will be evaluated by determining intraclass correlation coefficient (ICC) with 95% confidence interval, ranged between 0 and 1.

CONTACTS AND LOCATIONS:
Overall Officials: Betül Tepeli, Study Director — private balkan hospital
Locations (1):
- Betül Tepeli, Kırklareli, Lüleburgaz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] L'Insalata JC, Warren RF, Cohen SB, Altchek DW, Peterson MG. A self-administered questionnaire for assessment of symptoms and function of the shoulder. J Bone Joint Surg Am. 1997 May;79(5):738-48. PMID 9160947
- [Result] Vermeulen HM, Boonman DC, Schuller HM, Obermann WR, van Houwelingen HC, Rozing PM, Vliet Vlieland TP. Translation, adaptation and validation of the Shoulder Rating Questionnaire (SRQ) into the Dutch language. Clin Rehabil. 2005 May;19(3):300-11. doi: 10.1191/0269215505cr811oa. PMID 15859531
- [Result] Paul A, Lewis M, Shadforth MF, Croft PR, Van Der Windt DA, Hay EM. A comparison of four shoulder-specific questionnaires in primary care. Ann Rheum Dis. 2004 Oct;63(10):1293-9. doi: 10.1136/ard.2003.012088. PMID 15361390